CLINICAL TRIAL: NCT05529589
Title: Comparative Study of Anti-VEGF Effect and Visual Function in Vitreous Hemorrhage Patients With Diabetic Macular Edema After Pars Plana Vitrectomy With Inner Limiting Membrane Peeling or Not
Brief Title: Comparison of Restoration in Vitreous Hemorrhage Patients With DME After or Not Removing Inner Limiting Membrane
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: AVDME
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-08

CONDITIONS: Macular Edema Due to Diabetes Mellitus; Vitreous Hemorrhage
MeSH Terms: conditions — Vitreous Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Diabetic macular edema patient with inner limit membrane
- experimental group: Diabetic macular edema patient with inner limit membrane peeling

SUMMARY:
This study is conducted to compare the anti-VEGF effect and visual function in vitreous hemorrhage patients with diabetic macular edema after pars plana vitrectomy with inner limiting membrane peeling or not

ELIGIBILITY:
Inclusion Criteria:

* Patients with vitreous hemorrhage with diabetic macular edema and require vitreous surgery

Exclusion Criteria:

1. The patient's preoperative vitreous hemorrhage resulted in the failure of OCT to scan the macular region
2. The patient with a history of anti-VEGF therapy
3. Patients with DME in the contralateral eye requiring anti-VEGF therapy
4. Patients with contraindications of vitreous cavity resection
5. The patient has a history of intraocular surgery
6. The patient has active inflammatory disease
7. The patient has other retinal diseases that affect vision
8. The patient has other systemic diseases that required treatment with anti-VEGF drugs
9. Patient with contraindications to anti-VEGF therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with vitreous hemorrhage with DME who need vitreous surgery are of all ages and sexes
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-02-10 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Thickness change of retinal macular area | 12 months
  measurement of thickness of retinal macular area with macular optical coherence tomography after operation (0 day, 1 week, 1 months, 3 months, 6 months, 12 months)
Change of visual acuity | 12 months
  measurement of distance visual acuity with subjective refraction after operation (0 day, 1 week, 1 month, 3 months, 6 months, 12 months)

SECONDARY OUTCOMES:
Change of eye pressure | 12 months
  Measurement of contact tonometry with iCare TA01i tonometer after operation (0 day, 1 week, 1 month, 3 months, 6 months, 12 months)
B-mode ultrasound imaging | 12 months
  Existing or not of abnormal anatomical structure in posterior eye segment (0 day, 1 week, 1 month, 3 months, 6 months, 12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No